CLINICAL TRIAL: NCT04317092
Title: Multicenter Study on the Efficacy and Tolerability of Tocilizumab in the Treatment of Patients With COVID-19 Pneumonia
Brief Title: Tocilizumab in COVID-19 Pneumonia (TOCIVID-19)
Acronym: TOCIVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOCIVID-19; 2020-001110-38 (EudraCT Number)
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; pneumonia; tocilizumab; Interleukin-6
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: This is a multicenter, single-arm, open-label, phase 2 study. All the patients enrolled are treated with tocilizumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tocilizumab treatment (Experimental): All the patients enrolled are treated with tocilizumab.
  Interventions: Drug: Tocilizumab Injection

INTERVENTIONS:
Drug: Tocilizumab Injection — Tocilizumab 8 mg/kg (up to a maximum of 800mg per dose). A second administration (same dose) can be given after 12 hours if respiratory function has not recovered, at discretion of the Investigator.

SUMMARY:
This study project includes a single-arm phase 2 study and a parallel cohort study, enrolling patients with COVID-19 pneumonia.

DETAILED DESCRIPTION:
Phase 2 study: this is a multicenter, single-arm, open-label, phase 2 study. All the patients enrolled are treated with tocilizumab. Two-week (14 days) and one-month (30 days) lethality rates are the co-primary endpoints.

The parallel cohort includes patients who are treated with tocilizumab and cannot enter the phase 2 study because:

1. emergency conditions or infrastructural or operational limits prevented registration before the administration of the experimental drug or
2. they had been intubated more than 24 hours before registration or
3. the phase 2 study has been closed due to reached sample size.

This means that, after closure of the phase 2 enrolment, patients who might be eligible for the phase 2 study will be included in the observational cohort study.

The same information planned for the phase 2 cohort is required also for the parallel cohort study whose sample size is not defined a priori, and that will close at the end of the overall project. All the patients enrolled are treated with tocilizumab.

In both study groups (phase 2 and parallel cohort), participants receive one dose of Tocilizumab 8 mg/kg (up to a maximum of 800mg per dose). A second administration (same dose) can be given after 12 hours if respiratory function has not recovered, at discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender
2. No age limit
3. Informed consent for participation in the study (consent can be oral if a written consent cannot be expressed. If the subject is incapable of giving an informed consent and an authorized representative is not available without a delay that would, in the opinion of the Investigator, compromise the potential life-saving effect of the treatment this can be administered without consent. Consent to remain in the research should be sought as soon the conditions of the patient will allow it)
4. Virological diagnosis of SARS-CoV-2 infection (real-time PCR)
5. Hospitalized due to clinical/instrumental diagnosis of pneumonia
6. Oxygen saturation at rest in ambient air ≤93% or requiring oxygen therapy or mechanical ventilation either non invasive or invasive (intubated)
7. Patients with criteria #4 and #5 who have been already treated with tocilizumab before registration are eligible for the observational retrospective cohort

Exclusion Criteria:

1. Known hypersensitivity to tocilizumab or its excipients
2. Known active infections or other clinical condition that contraindicate tocilizumab and cannot be treated or solved according to the judgement of the clinician
3. ALT / AST> 5 times the upper limit of the normality
4. Neutrophils <500 / mmc
5. Platelets <50.000 / mmc
6. Bowel diverticulitis or perforation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2023-12-19 (Estimated); Study Completion 2023-12-19 (Estimated)

PRIMARY OUTCOMES:
Lethality rate two weeks after registration | up to 15 days
  2-week lethality is defined as the ratio of the number of subjects dead within 14 days from study start out of phase 2 patients with baseline information.
Lethality rate one month after registration | up to 1 month
  1-month lethality is defined as the ratio of the number of subjects dead within 30 days from study start out of phase 2 patients with baseline information.

SECONDARY OUTCOMES:
Interleukin-6 level | baseline, during treatment (cycle 1 and 2 every 12 hours) up to 1 month
  IL-6 levels will be assessed using commercial ELISA method.
Lymphocyte count | baseline, during treatment (cycle 1 and 2 every 12 hours) up to 1 month
  Lymphocyte count assessed by routinely used determination of blood count
CRP (C-reactive protein) level | baseline, during treatment (cycle 1 and 2 every 12 hours) up to 1 month
  CRP is assessed by routinely used determination of CRP
PaO2 (partial pressure of oxygen) / FiO2 (fraction of inspired oxygen, FiO2) ratio (or P/F ratio) | baseline, during treatment (cycle 1 and 2 every 12 hours) up to 1 month
  calculated from arterial blood gas analyses (values from 300 to 100)
Change of the SOFA (Sequential Organ Failure Assessment) | baseline, during treatment (cycle 1 and 2 every 12 hours) up to 1 month
  It evaluates 6 variables, each representing an organ system (one for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems), and scored from 0 (normal) to 4 (high degree of dysfunction/failure). Thus, the maximum score may range from 0 to 24.
Number of participants with treatment-related side effects as assessed by Common Terminology Criteria for Adverse Event (CTCAE) version 5.0 | during treatment and up to 30 days after the last treatment dose
  graded according to CTCAE citeria (v5.0)
Radiological response | at baseline (optional), after seven days and if clinically indicated (up to 1 month)
  Thoracic CT scan or Chest XR
Duration of hospitalization | from baseline up to patient's discharge (up to 1 month)
  Days of hospitalization
Remission of respiratory symptoms | up to 1 month
  time to invasive mechanical ventilation (if not previously initiated) calculated from baseline to intubation
Remission of respiratory symptoms | up to 1 month
  time to definitive extubation calculated from intubation (any time occurred) to extubation in days
Remission of respiratory symptoms | up to 1 month
  time to independence from non-invasive mechanical ventilation calculated in days
Remission of respiratory symptoms | up to 1 month
  time to independence from oxygen therapy in days

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Perrone, MD, PhD, Principal Investigator — Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale
Locations (27):
- Italy (27):
  - Azienda Ospedaliera "SS. Antonio e Biagio e C. Arrigo" (Dipartimento Internistico SSD Reumatologia), Alessandria
  - Ospedale di Busto Arsizio ASST Valle Olona (U.O.C. Malattie Infettive), Busto Arsizio
  - A.O.U. Policlinico V. Emanuele (U.O. di Malattie infettive, U.O. di Anestesia e Rianimazione, U.O. di Medicina d'Urgenza), Catania
  - AOE Cannizzaro di Catania (U.O. di Malattie Infettive, U.O. di Anestesia e Rianimazione, U.O., Catania
  - Ospedale Annunziata Azienda Ospedaliera di Cosenza (U.O.C. Malattie Infettive), Cosenza
  - ASST OVEST MILANESE presidi Legnano - Magenta, Magenta
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - A.O.U. di Modena (Dipartimento Chirurgie Generali e Specialità Chirurgiche - Struttura Complessa di Anestesia e Rianimazione I), Modena
  - A.O.U. di Modena (Dipartimento Chirurgie Generali e Specialità Chirurgiche - Struttura Complessa di Anestesia e Rianimazione II), Modena
  - A.O.U. di Modena (Dipartimento Medicine Specialistiche - Struttura Complessa Malattie Infettive), Modena
  - Dipartimento Medicine Specialistiche - Struttura Complessa Malattie dell'Apparato Respiratorio, Modena
  - A.O.R.N. Ospedale dei Colli Monaldi-Cotugno-CTO (U.O.C. Oncologia), Naples
  - National Cancer Institute, Naples
  - A.O.R.N. Ospedale dei Colli Monaldi-Cotugno-CTO (U.O.C. Anestesia Rianimazione e terapia intensiva), Naples
  - A.O.R.N. Ospedale dei Colli Monaldi-Cotugno-CTO (U.O.C. Malattie Infettive ad indirizzo respiratorio), Naples
  - A.O. Ospedali Riuniti Marche Nord - Presidio Ospedaliero San Salvatore di Pesaro (UOC Pronto Soccorso e Medicina d'Urgenza), Pesaro
  - Denominazione: UOC di Medicina e Chirurgia d'Accettazione e d'Urgenza dell'Ospedale Santa Maria delle Grazie di Pozzuoli, Pozzuoli
  - Ospedale Santa Maria delle Croci, AUSL della Romagna (U.O. Anestesia e Rianimazione), Ravenna
  - Grande Ospedale Metropolitano, Reggio Calabria, Reggio Calabria
  - Ospedale Infermi, AUSL della Romagna (U.O. Malattie Infettive), Rimini
  - Policlinico Gemelli (U.O.C. Dipartimento Scienze di Laboratorio e Infettivologiche), Rome
  - ASST Sette Laghi (Dipartimento di Medicina Interna), Varese
  - ASST Sette Laghi (Dipartimento Emergenze ed Urgenze), Varese
  - ASST Sette Laghi (U.O.C. Anestesia e Rianimazione Neurochirurgica e Generale), Varese
  - ASST Sette Laghi (U.O.C. Malattie Infettive e Tropicali), Varese
  - A.O.U. Integrata di Verona (Dip. Malattie Infettive), Verona
  - Ospedale Magalini (U.O. Malattie Infettive), Villafranca di Verona

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request to the Principal Investigator of the study
  The following IPD will be available for sharing:
  1. Baseline characteristics of patients
  2. Treatment data
  3. Safety data
  4. Follow-up data
Supporting Information: Study Protocol, SAP
Time Frame: After peer-reviewed publication of the primary results, with no time limits
Access Criteria: Motivated requests to access to IPD are to be sent by email to the Principal Investigator (f.perrone@istitutotumori.na.it)

REFERENCES:
- [Derived] Perrone F, Piccirillo MC, Ascierto PA, Salvarani C, Parrella R, Marata AM, Popoli P, Ferraris L, Marrocco-Trischitta MM, Ripamonti D, Binda F, Bonfanti P, Squillace N, Castelli F, Muiesan ML, Lichtner M, Calzetti C, Salerno ND, Atripaldi L, Cascella M, Costantini M, Dolci G, Facciolongo NC, Fraganza F, Massari M, Montesarchio V, Mussini C, Negri EA, Botti G, Cardone C, Gargiulo P, Gravina A, Schettino C, Arenare L, Chiodini P, Gallo C; TOCIVID-19 investigators, Italy. Tocilizumab for patients with COVID-19 pneumonia. The single-arm TOCIVID-19 prospective trial. J Transl Med. 2020 Oct 21;18(1):405. doi: 10.1186/s12967-020-02573-9. PMID 33087150
- [Derived] Chiodini P, Arenare L, Piccirillo MC, Perrone F, Gallo C. A phase 2, open label, multicenter, single arm study of tocilizumab on the efficacy and tolerability of tocilizumab in the treatment of patients with COVID-19 pneumonia (TOCIVID-19 trial): Statistical analysis plan. Contemp Clin Trials Commun. 2020 Dec;20:100665. doi: 10.1016/j.conctc.2020.100665. Epub 2020 Oct 7. PMID 33043164
- [Derived] Piccirillo MC, Ascierto P, Atripaldi L, Cascella M, Costantini M, Dolci G, Facciolongo N, Fraganza F, Marata A, Massari M, Montesarchio V, Mussini C, Negri EA, Parrella R, Popoli P, Botti G, Arenare L, Chiodini P, Gallo C, Salvarani C, Perrone F. TOCIVID-19 - A multicenter study on the efficacy and tolerability of tocilizumab in the treatment of patients with COVID-19 pneumonia. Study protocol. Contemp Clin Trials. 2020 Nov;98:106165. doi: 10.1016/j.cct.2020.106165. Epub 2020 Oct 6. PMID 33031955